CLINICAL TRIAL: NCT03293784
Title: TNF-Inhibitor as Immune Checkpoint Inhibitor for Advanced MELanoma - A Phase Ib Clinical Study
Brief Title: TNF-Inhibitor as Immune Checkpoint Inhibitor for Advanced MELanoma
Acronym: TICIMEL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16CUTA07
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Melanoma
Keywords: Melanoma; Immune checkpoint; Nivolumab; Ipilimumab; Infliximab; Certolizumab; PD-1; TNFa; CTLA-4
MeSH Terms: conditions — Melanoma; Diabetes Mellitus, Insulin-Dependent, 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COHORT 1 (Other): Nivolumab+Ipilimumab in combination with Anti TNF-α Certolizumab
  Interventions: Combination Product: Nivolumab+Ipilimumab in combination with Anti TNF-α Certolizumab
- COHORT 2 (Other): Nivolumab+Ipilimumab in combination with Anti TNF-α Infliximab
  Interventions: Combination Product: Nivolumab+Ipilimumab in combination with Anti TNF-α Infliximab

INTERVENTIONS:
Combination Product: Nivolumab+Ipilimumab in combination with Anti TNF-α Certolizumab — Induction phase: Nivolumab (1mg/kg) and Ipilimumab (3 mg/kg) injected at Week 0, 3, 6, and 9 with Certolizumab injected at the dose of 400mg at weeks 0, 3, and 6, and at the dose of 200mg at week 9.
  Maintenance phase: Nivolumab (3 mg/kg) alone injected from week 12 and then every 2 weeks with Certolizumab (200 mg) injected from week 12 and then every 2 weeks.
  Arms: COHORT 1
Combination Product: Nivolumab+Ipilimumab in combination with Anti TNF-α Infliximab — Induction phase: Nivolumab (1mg/kg) and Ipilimumab 3 mg/kg injected at Week 0, 3, 6, and 9 with Infliximab (5mg/kg) injected at weeks 0, 3 and 6.
  Maintenance phase: Nivolumab (3 mg/kg) alone injected from week 12 and then every 2 weeks with Infliximab (5mg/kg) injected from week 14 and then every 8 weeks.
  Arms: COHORT 2

SUMMARY:
This is a Phase 1b, open-label study of immune checkpoints inhibitors Nivolumab+Ipilimumab administered in combination with the anti-TNF-α either Infliximab or Certolizumab, in patients with advanced melanoma.

DETAILED DESCRIPTION:
The study will be conducted in 2 consecutive parts:

* Part 1 with 2 parallel cohorts (Nivolumab+Ipilimumab administered in combination with anti-TNF-α Certolizumab (Cohort 1) and Nivolumab+Ipilimumab administered in combination with anti-TNF-α Infliximab (Cohort 2)). 6 patients will be included in each cohort.
* Part 2 (expansion phase) will then be scheduled after the most promising combination has been confirmed; the choice of the combination will be based on safety, efficacy, and PD data observed in both cohorts during the Part 1 of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologically-proven metastatic and/or unresectable melanoma (stage IIIc-IV, M1a-c as per AJCC 2009), including mucosal melanoma, without evidence of active intra-cranial disease.
2. Subjects are included regardless of BRAFV600 mutation status. BRAFV600 mutation status must be documented.
3. Measurable disease per RECIST 1.1
4. Age ≥18 years and ≤70 years at the time of study entry.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
6. Life expectancy of at least 3 months.
7. Patient able to participate and willing to give informed consent prior to performance of any study-related procedures and to comply with the study protocol.
8. Screening laboratory values must meet the following criteria and should be obtained prior to commencement of treatment:

   White blood count (WBC) ≥ 2000/μL Neutrophils ≥ 1500/μL Platelets ≥ 100 x103/μL Hemoglobin > 9.0 g/dL

   Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

   Female CrCl = (140 - age in years) x weight in kg x 0.85 / 72 x serum creatinine in mg/dL Male CrCl = (140 - age in years) x weight in kg x 1.00 / 72 x serum creatinine in mg/dL AST/ALT ≤ 3 x ULN (except subjects with hepatic metastasis, who can have AST/ALT ≤ 5 x ULN) Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
9. Adequate cardiac and respiratory functions defined as New York Heart Association (NYHA) class 1 and SaO2 > 90%.
10. Patient must be naïve to systemic treatment for locally advanced and/or metastatic disease (i.e., no prior systemic anticancer therapy for advanced disease; stage IIIc and IV). Prior adjuvant therapies (including Interferon α and Ipilimumab) is permitted if it was completed at least 12 weeks before start of treatment and all related AEs have either returned to baseline or stabilized.
11. Prior radiotherapy or radiosurgery must have been completed at least 4 weeks prior to the first dose of the study treatment.
12. Women of childbearing potential (WOCBP) must use two appropriate methods of contraception to avoid pregnancy for 23 weeks (30 days plus the time required for Nivolumab/Ipilimumab to undergo five half-lives) after the last dose of investigational drug.
13. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment.
14. Men who are sexually active with WOCBP must use two contraceptive methods including at least one method with a failure rate of less than 1% per year for a period of 31 weeks after the last dose of investigational product. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception.
15. Absence of any psychological, familial, sociological or geographical condition that potentially hampers compliance with the study protocol and follow-up after treatment discontinuation schedule.
16. Patient affiliated to a Social Health Insurance in France.
17. Patient must provide written informed consent prior to any study specific procedures.

Exclusion Criteria:

1. Patient pregnant, or breast-feeding.
2. Uveal melanoma.
3. Active and/or symptomatic intra cranial metastasis (including melanomatous meningitis). Patients with intra cranial metastasis may be eligible if all known lesions have been treated with stereotactic radiotherapy or surgery or both AND there has been no magnetic resonance imaging (MRI) evidence of disease progression in the CNS for ≥ 4 weeks after treatment and within 28 days prior the first dose of study drug administration.
4. Previous treatment with B-RAF or MEK inhibitors within 12 weeks prior start of treatment.
5. Hypersensitivity to the drugs of the study.
6. Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
7. Clinically significant cardiac dysfunction including congenital, familial, and genetic cardiac disorders, current instable angina, current symptomatic congestive heart failure of NYHA class 2 and higher, current uncontrolled hypertension ≥ grade 3; Left Ventricular Ejection Fraction (LVEF) below institutional lower limit of normal (LLN) or below 50%, whichever is lower.
8. Patient with active malignancy other than melanoma or a history of previous within the past 3 years; except for patients with resected Basal cell carcinoma or resected Spindle cell carcinoma, resected carcinoma in situ of the cervix and resected carcinoma in situ of the breast.
9. History of untreated tuberculosis and/or positive quantiferon test without previous prophylaxis tuberculosis treatment, or untreated active infection with mycobacterium tuberculosis. For patients with asymptomatic (including radiologic symptoms) infection with mycobacterium tuberculosis, inclusion may be possible after 4 weeks of adequate antibiotics treatment.
10. Active, known or suspected autoimmune disease including but not restricted to multiple sclerosis, optical nevritis and demyelinating neuropathy. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
11. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus (HCV ribonucleic acid or HCV antibody) indicating acute or chronic infection.
12. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
13. Vaccination with any live attenuated conventional vaccine within the 3 months preceding the start of study treatment.
14. Any current severe or uncontrolled disease, including, but not limited to ongoing or active infection.
15. Patient included in another study with an experimental molecule and/or procedure.
16. Unwillingness or inability to provide written informed consent.
17. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the compliance of treatment and the study protocol.
18. Patient who has forfeited his/her freedom by administrative or legal award or who is under guardianship.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) incidence, in part 1 of the study. | 12 weeks per patient (part 1)
  For each patient, DLT incidence will be evaluated during the Part 1 of the study: 12 weeks after the initial dose of study drug.

SECONDARY OUTCOMES:
Safety and tolerability according to the classification of the National Cancer Institute Common Toxicity Criteria for Adverse Effects (NCI-CTCAE) Version 4.03. | 15 months per patient
  The assessment of safety and tolerability will be based on the incidence of Adverse Events (AEs), Serious Adverse Events, AEs leading to discontinuation, and death. In addition, clinical laboratory test abnormalities will be examined. Tolerability will be evaluated by collecting dose interruptions and dose delays.
Progression Free Survival | 24 months per patient
  Progression Free Survival (PFS) is defined as the time from inclusion until progression or deaths; patients alive at last follow-up news are censored at this date.
Objective Response Rate | 24 months per patient
  Objective Response Rate (ORR) is defined as the number of patients with Best Overall Response divided by the number of included patients in each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MEYER, Principal Investigator — Institut Claudius Regaud
Locations (1):
- Institut Claudius Regaud IUCT-ONCOPOLE, Toulouse, France

REFERENCES:
- [Derived] Montfort A, Filleron T, Virazels M, Dufau C, Milhes J, Pages C, Olivier P, Ayyoub M, Mounier M, Lusque A, Brayer S, Delord JP, Andrieu-Abadie N, Levade T, Colacios C, Segui B, Meyer N. Combining Nivolumab and Ipilimumab with Infliximab or Certolizumab in Patients with Advanced Melanoma: First Results of a Phase Ib Clinical Trial. Clin Cancer Res. 2021 Feb 15;27(4):1037-1047. doi: 10.1158/1078-0432.CCR-20-3449. Epub 2020 Dec 3. PMID 33272982